CLINICAL TRIAL: NCT03593668
Title: Effect and Safety of Benaglutide or Metformin in Patients With Simple Obesity Who Have Inadequate Weight Control :A Randomized, Open, Controlled and Single-site Clinical Trail
Brief Title: Effect and Safety of Benaglutide or Metformin in Patients With Simple Obesity Who Have Inadequate Weight Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET2018
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Obesity; Drug
Keywords: Metformin; Benaglutide
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Metformin Hydrochloride Tablet 500mg po by month,three times a day for 12 weeks
  Interventions: Drug: Metformin
- Benaglutide (Active Comparator): Benaglutide Injection 0.2mg, iH,po, three times a day for 3 12 weeks
  Interventions: Drug: Benaglutide

INTERVENTIONS:
Drug: Metformin — 2-week dose adjustment period（0-2weeks）[before meals] 0-2d： - ;250mg，po; -. 3-4d： - ;250mg，po; 250mg，po. 5-6d： 250mg，po; 250mg，po; 250mg，po. 7-9d: 250mg，po; 500mg，po; 250mg，po. 10-11d: 250mg，po; 500mg，po; 500mg，po. 12-14d: 500mg，po; 500mg，po; 500mg，po.
  10-week dose stabilization period（3-12weeks） Metformin Hydrochloride Tablet 500mg tid po.
  Other Names: Glucophage; Metformin Hydrochloride Tablet
  Arms: Metformin
Drug: Benaglutide — 2-week dose adjustment period（0-2weeks） [before meals] 0-2d: -; 0.1mg，iH; -; 3-4d: -; 0.1mg，iH; 0.1mg，iH; 5-6d: 0.1mg，iH; 0.1mg，iH; 0.1mg，iH; 7-9d: 0.1mg，iH; 0.2mg，iH; 0.1mg，iH; 10-11d: 0.1mg，iH; 0.2mg，iH; 0.2mg，iH; 12-14d: 0.2mg，iH; 0.2mg，iH; 0.2mg，iH.
  10-week dose stabilization period（3-12weeks） Benaglutide Injection 0.2mg，100ul，tid，iH
  Other Names: Benaglutide Injection
  Arms: Benaglutide

SUMMARY:
This is a randomized, open, controlled and single-site clinical trail to investigate the effect and safety of Benaglutide or Metformin in patients with simple obesity who have inadequate weight control.

DETAILED DESCRIPTION:
This is a randomized, open, controlled and single-site clinical trail to investigate the effect and safety of Benaglutide or Metformin in patients with simple obesity who have inadequate weight control.

Screening will be made to select eligible participants before intervention. Patients were randomly assigned to one of two groups(metformin or benaglutide) for therapies for 12 weeks including a two-week dose adjustment period and a 10-week dose stabilization period. Lifestyle interventions will be maintained during the treatment period. Subjects are followed up every 4 weeks for examinations.At the end of the study, data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

(1)20 years old≤70 years old; (2) simple obesity, gender is not limited; (3) 28.0≤BMI≤37.5kg/m2; (4) Before the screening period, the body weight was controlled by lifestyle interventions (diet and exercise) for at least 3 months, and weight was decreased by <5% from baseline; (5) Agree to sign the informed consent form;

Exclusion Criteria:

1. Accurately diagnosed as having type 1 or type 2 diabetes according to the WHO 1999 diagnostic criteria;
2. Use weight loss drugs within 3 months before screening;
3. Metformin was used within the first 3 months of screening;
4. Malignant tumors (excluding basal cell or squamous cell carcinoma treated) within 5 years before enrollment
5. Alanine aminotransferase or aspartate aminotransferase > 3 times the upper limit of normal or total serum bilirubin (TB) >34.2 μmol/L (>2 mg/dL)
6. Patients with moderate/severe renal impairment or end-stage renal disease (eGFR < 60 mL/min/1.73 m2); male subjects with serum creatinine (Cr) ≥133 μmol/L (≥1.50 mg/dL Serum Cr in female subjects was ≥124 μmol/L (>1.40 mg/dL);
7. Severe heart, lung, nervous, mental and infectious diseases;
8. Pregnancy, lactation and recent pregnancy plans;
9. Alternate or chronic systemic corticosteroid therapy, defined as treatment with any dose of systemic corticosteroids within 3 months of enrollment visit V1 > 4 weeks
10. History of alcohol abuse, history of abuse of active drugs (opioids, analgesics, etc.) within 6 months before enrollment;
11. Give any other test drug within 30 days before enrollment or within 5 half-lives of other test drugs;
12. Patients with past history or family history of medullitary thyroid cancer (MTC) and patients with type 2 multiple endocrine tumor syndrome (MEN2);
13. Inability to tolerate benalutide, metformin;
14. Any influence of the investigator's judgment on enrollment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-30 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | Change from Baseline after 12 weeks treatment
  Changes in body weight from baseline were observed in patients with simple obesity after 12 weeks of treatment intervention.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) of subjects | Change from Baseline after 12 weeks treatment
  All 30 subjects of each group would be evaluted by changes in body mass index (BMI) after 12 weeks treatment
Changes in Body Fat Levels | Change from Baseline after 12 weeks treatment
  Changes in Body Fat Levels from Baseline: Body Composition Analysis
Changes in blood lipid levels | Change from Baseline after 12 weeks treatment
  The changes in blood lipid levels such as cholesterol, triglycerides, low-density lipoprotein, high-density lipoprotein will be measured at the beginning and the end.

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China